CLINICAL TRIAL: NCT00388466
Title: Cystic Fibrosis: Improvement of Muscle Force and Function by Whole Body Vibration Exercise
Brief Title: Whole Body Vibration - a New Therapeutic Approach to Improve Muscle Function in CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-005
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2006-10-16 (Estimated); Status verified 2006-10

CONDITIONS: Cystic Fibrosis
Keywords: whole body vibration; muscle function; cystic fibrosis; mechanography; chair-rising-test
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Device: GALILEO

SUMMARY:
The purpose of this study is to evaluate the effects of whole body vibration (WBV) on muscle function in adult CF-patients.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is the most common chronic hereditary disease in Caucasians. Due to improved therapy and better understanding of the disease, life expectancy has risen to an average of 38 years and is continuing to rise. With the increased life-expectancy it becomes even more important to maintain functional activity as part of quality of life. Mechanical stimulation in form of whole body vibration (WBV) is a new type of exercise currently tested in sports, geriatrics and rehabilitation. It has recently been found to be a safe and efficient method to activate muscular activity via stretch reflexes leading to improvement of muscular performance, body balance and physical functioning.

10 patients of the CF Center Cologne, Germany, took part in the Galileo study. They were provided by the vibrating platform (Galileo 2000)for whole body vibration training at home. The patients were standing in an upright position receiving vertical vibration of frequencies between 20-25 Hz. This vibration exercise evokes muscle contractions via stretch reflexes improving muscular activity. The training schedule consisted of three 3-minute sessions twice a day 5 days per week for 3 months.

Every 4 weeks the patients were seen for assessment of muscle function to evaluate the effects of this new intervention.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Cystic Fibrosis
* age older than 18 years

Exclusion Criteria:

* hypersplenic syndrome
* acute arthritis or osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-06; Study Completion 2006-08

PRIMARY OUTCOMES:
muscle force at the beginning of the study and after 3 months
muscle power at the beginning of the study and after 3 months

SECONDARY OUTCOMES:
pulmonary function testing at the beginning of the study and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Schoenau, Prof., Study Chair — University Children´s Hospital Cologne, Germany
Locations (1):
- CF Center Cologne, University Children's Hospital, Cologne, Germany

REFERENCES:
- [Background] Fricke O, Weidler J, Tutlewski B, Schoenau E. Mechanography--a new device for the assessment of muscle function in pediatrics. Pediatr Res. 2006 Jan;59(1):46-9. doi: 10.1203/01.pdr.0000191580.07644.1c. Epub 2005 Dec 2. PMID 16327004